CLINICAL TRIAL: NCT05061251
Title: An Open-Label Surgical Window of Opportunity Study Evaluating Pharmacodynamic Response of Orally Administered BAY 2402234 in Subjects With Recurrent Glioma, IDH Mutant, Grade 3 or 4
Brief Title: Surgical Window of Opportunity Study of Orally Administered BAY 2402234 in Recurrent Glioma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Drug availability
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Kalil Abdullah, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAY 2402234
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Glioma; IDH Mutation
MeSH Terms: conditions — Glioma | interventions — orludodstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- BAY 2402234 (Experimental): Patients will receive 1 dose (5mg) orally, per day of BAY 2402234 for the 2 days prior to standard-of-care craniotomy for tumor resection and 1 dose on the morning of surgery, for a total of 3 administered doses.
  Interventions: Drug: BAY 2402234

INTERVENTIONS:
Drug: BAY 2402234 — Patients will receive 3 doses of 5mg each of BAY 2402234. Drug will be given Day 1 and Day 2 prior to standard-of-care craniotomy for tumor resection and 1 dose on the morning of surgery.

SUMMARY:
This study aims to look at how BAY 2402234 responds in body in patients with recurrent glioma.

DETAILED DESCRIPTION:
To characterize the biological activity of BAY 2402234 in recurrent glioma, IDH-mutant, Grade 3/4 using liquid chromatography-mass spectrometry (LC-MS). The tissue orotate:carbamoyl aspartate ratio will serve as the primary pharmacodynamic biomarker and will be characterized via LC-MS.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Histologically and/or genomically documented recurrent or progressive astrocytoma, IDH-mutant, grade 3 or 4 (diagnosis established by the presence of an IDH1 or IDH2 mutation along with grade 3 or 4 radiographic findings)
* Interval of at least 12 weeks from completion of adjuvant radiotherapy for gliomas to dosing, or surgical confirmation of recurrent disease
* Performance status measured via Karnofsky Performance Score of ≥ 60
* Confirmed measurable disease per response assessment in neuro-oncology criteria (RANO)
* Participants should have at least one 1.5cm x 1.5cm region of enhancing and non-enhancing tumor within the surgically accessible region
* Ability of neurosurgeon to resect tumor
* Laboratory values at the Screening Visit:

  * ANC count ≥1,500/mm3;
  * Platelets ≥150,000/mm3;
  * Hemoglobin > 9g/dL
  * Total bilirubin ≤1.5 × the upper limit of normal (ULN) (subjects with Gilbert's Syndrome are allowed if direct bilirubin is within normal limits)
  * Aspartate aminotransferase (AST [SGOT]) ≤3× the ULN
  * Alanine aminotransferase (ALT [SGPT]) ≤3 × the ULN
  * Serum creatinine ≤1.5 mg/dL or a calculated creatinine clearance ≤60 mL/min
  * Negative serum B-hCG test in women of childbearing potential (defined as women ≤50 years of age, or >50 years of age with a history of amenorrhea for ≤12 months prior to study entry)
* All men, as well as women of child-bearing potential must agree to use dual contraceptive methods (hormonal or barrier method of birth control; abstinence) while on the study drug and for 3 months afterward. Men must also refrain from sperm donation for 4 months after treatment with BAY 2402234. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Patients under age 18 (due to fundamental difference between pediatric and adult gliomas)
* Treatment with an IDH inhibitor within 90 days of enrollment
* Treatment with temozolomide less than 23 days from study initiation, treatment with CCNU or BCNU less than 42 days from study initiation, or treatment with any cancer-directed systemic therapy less than 4 weeks or 5 half-lives from study initiation, whichever is shorter
* Any immunomodulatory drug or molecularly targeted, monoclonal antibody, within 14 days prior to initiation of study drug
* Use of any investigational agents within 28 days of baseline or 5 half-lives from study initiation, whichever is shorter
* Increasing corticosteroid requirement or a dose of >24mg per day of dexamethasone or an equivalent dose of other corticosteroids for longer than 48 hours within 7 days prior to study initiation
* Radiotherapy within 12 weeks prior to registration unless surgical confirmation of recurrent disease
* Presence of an acute or chronic toxicity of prior chemotherapy, with the exception of alopecia or lymphopenia, that has not resolved to ≤ Grade 1, as determined by National Cancer Institute CTCAE v5.0
* Major surgery within 28 days prior to initiation of study drug
* Active or clinically unstable bacterial, viral, or fungal infection requiring systemic therapy
* Known human immunodeficiency virus or acquired immunodeficiency syndrome-related illness
* Any of the following within 6 months prior to initiation of study drug: uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary or peripheral artery bypass graft surgery, transient ischemic attack
* Pulmonary embolism within 1 month prior to initiation of study drug
* Unstable cardiac dysrhythmias or persistent prolongation of the QTc interval to >450 msec for males or >470 msec for females
* Any contraindication to contrast-enhanced MRI examination
* Evidence of clinically significant intracranial hemorrhage
* Previous history of an additional emergency, except for non-squamous-cell carcinoma of skin or carcinoma-in-situ of the uterine cervix, unless the tumor was treated with curative intent more than 2 years prior to study entry
* Requires anti-seizure medications that are known to be strong inducers of CYP3A4/5 enzymes (carbamazepine, phenobarbital, phenytoin). Strong inhibitors and/or strong inducers of CYP3A4 should not be administered within 14 days or 5 half-lives (whichever is shorter) of the start of BAY 2402234 treatment, or during BAY 2402234 treatment, unless there is an emergent or life-threatening medical condition
* Pregnant or lactating female
* Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study
* Difficulty swallowing or malabsorption syndrome; refractory nausea & vomiting, chronic gastrointestinal disease or previous significant bowel resection with clinically significant sequelae that would preclude adequate absorption of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Biological activity of BAY 2402234 | 3 days up tp day of surgery
  The primary endpoint is to characterize the biological activity of BAY 2402234 using liquid chromatography-mass spectrometry (LC-MS). The tissue orotate:carbamoyl aspartate ratio will serve as the primary pharmacodynamic biomarker and will be characterized via LC-MS.

SECONDARY OUTCOMES:
Adverse Event Monitoring | 28 days after the final administered dose of BAY 2402234
  To monitor adverse events during treatment with BAY 2402234 and document them in accordance with the Common Technology Criteria for Adverse Events (CTCAE) Version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Kalil g Abdullah, MD, MSc, Principal Investigator — UT Southwestern/ Simmons CC